CLINICAL TRIAL: NCT01684878
Title: A Two-Part, Randomized Phase III, Double-Blind, Multicenter Trial Assessing The Efficacy And Safety of Pertuzumab In Combination With Standard Chemotherapy Vs. Placebo Plus Standard Chemotherapy In Women With Recurrent Platinum-Resistant Epithelial Ovarian Cancer And Low HER3 mRNA Expression
Brief Title: Pertuzumab in Platinum-Resistant Low Human Epidermal Growth Factor Receptor 3 (HER3) Messenger Ribonucleic Acid (mRNA) Epithelial Ovarian Cancer (PENELOPE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MO28113; 2011-005975-17 (EudraCT Number)
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Gemcitabine; Drug Therapy; Paclitaxel; pertuzumab; Topotecan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Part 1: Pertuzumab + Topotecan (Experimental): Participants received pertuzumab and topotecan in cycles of 3 weeks until progressive disease as per investigator's assessment, unacceptable toxicity, withdrawal of consent, or death.
  Interventions: Drug: Paclitaxel (Chemotherapy); Drug: Pertuzumab; Drug: Topotecan (Chemotherapy)
- Part 1: Pertuzumab + Paclitaxel (Experimental): Participants received pertuzumab and paclitaxel in cycles of 3 weeks until progressive disease as per investigator's assessment, unacceptable toxicity, withdrawal of consent, or death.
  Interventions: Drug: Paclitaxel (Chemotherapy); Drug: Pertuzumab; Drug: Placebo
- Part 2: Pertuzumab+Chemotherapy (Experimental): Participants received pertuzumab and chemotherapy (paclitaxel or topotecan or gemcitabine) in cycles of 3 weeks until progressive disease as per investigator's assessment, unacceptable toxicity, withdrawal of consent, or death. Chemotherapy was administered as per investigators discretion.
  Interventions: Drug: Gemcitabine (Chemotherapy); Drug: Paclitaxel (Chemotherapy); Drug: Pertuzumab; Drug: Topotecan (Chemotherapy)
- Part 2: Placebo+Chemotherapy (Placebo Comparator): Participants received pertuzumab matching placebo and chemotherapy (paclitaxel or topotecan or gemcitabine) in cycles of 3 weeks until progressive disease as per investigator's assessment, unacceptable toxicity, withdrawal of consent, or death. Chemotherapy was administered as per investigators discretion.
  Interventions: Drug: Gemcitabine (Chemotherapy); Drug: Paclitaxel (Chemotherapy); Drug: Placebo; Drug: Topotecan (Chemotherapy)

INTERVENTIONS:
Drug: Gemcitabine (Chemotherapy) — Participants administered gemcitabine at a dosage of 1000 milligrams per square meter (mg/m^2) intravenous (IV) infusion on Days 1 and 8 every 3 weeks.
  Arms: Part 2: Pertuzumab+Chemotherapy; Part 2: Placebo+Chemotherapy
Drug: Paclitaxel (Chemotherapy) — Participants administered paclitaxel at a dosage of 80 mg/m^2 as 1 hour IV infusion on Days 1, 8 and 15 every 3 weeks.
Drug: Pertuzumab — Participants administered pertuzumab 840 milligrams (mg) IV infusion on Day 1 of the first treatment cycle as a loading dose, followed by 420 mg on Day 1 of each subsequent 3 weekly cycle.
  Arms: Part 1: Pertuzumab + Paclitaxel; Part 1: Pertuzumab + Topotecan; Part 2: Pertuzumab+Chemotherapy
Drug: Placebo — Participants administered pertuzumab matching placebo IV infusion on Day 1 of each 3 weekly cycle.
  Arms: Part 1: Pertuzumab + Paclitaxel; Part 2: Placebo+Chemotherapy
Drug: Topotecan (Chemotherapy) — Participants administered topotecan at a dosage of 1.25 mg/m^2 as a 30 minute IV infusion daily on Days 1 to 5 every 3 weeks.
  Arms: Part 1: Pertuzumab + Topotecan; Part 2: Pertuzumab+Chemotherapy; Part 2: Placebo+Chemotherapy

SUMMARY:
This two-part, multicenter study will evaluate the safety, tolerability and efficacy of pertuzumab in combination with standard chemotherapy in women with recurrent platinum-resistant epithelial ovarian cancer. In the non-randomized Part 1 safety run-in, participants will receive pertuzumab plus either topotecan or paclitaxel. In the randomized, double-blind Part 2 of the study, participants will receive either pertuzumab or placebo in combination with chemotherapy (topotecan, paclitaxel, or gemcitabine).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed epithelial ovarian, primary peritoneal, and/or fallopian tube cancer that is platinum-resistant or refractory
* Low Human epidermal growth factor receptor (HER) 3 messenger ribonucleic acid (mRNA) expression
* At least one measurable and/or non-measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version (V) 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Left ventricular ejection fraction (LVEF) greater than or equal to (>/=) 50 percent (%)
* Negative serum pregnancy test in women of childbearing potential
* Women of childbearing potential must agree to use effective contraception as defined by protocol during and for at least 6 months post study treatment

Exclusion Criteria:

* Non-epithelial tumors
* Ovarian tumors with low malignant potential (borderline tumors)
* History of other malignancy of prognostic relevance within the last 5 years, except for carcinoma in situ of the cervix or basal cell carcinoma, or tumors with a negligible risk for metastasis or death, such as adequately controlled basal-cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or carcinoma in situ of the breast
* Previous treatment with more than 2 chemotherapy regimens
* Any prior radiotherapy to the pelvis or abdomen
* History or evidence on physical/neurological examination of central nervous system disease unrelated to cancer (uncontrolled seizures), unless adequately treated with standard medical therapy
* Pre-existing peripheral neuropathy >/= common toxicity criteria (CTC) grade 2 (applicable for paclitaxel cohort only)
* Inadequate organ function
* Uncontrolled hypertension or clinically significant cardiovascular disease
* Current known infection with human immunodeficiency virus (HIV) or active infection with hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Current chronic daily treatment with corticosteroids (>/= 10 mg per day of methylprednisolone or equivalent), excluding inhaled steroids
* History of receiving any investigational treatment within 28 days prior to first study drug administration
* For Part 2 of the trial: prior enrollment into Part 1 of the trial
* Concurrent participation in any therapeutic clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2012-10-22 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2016-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (68):
- Austria (2):
  - Tiroler Landeskrankenanstalten Ges.M.B.H.; Abt. Für Gynäkologie, Innsbruck
  - Medizinische Universität Wien; Univ.Klinik für Frauenheilkunde - Klinik für Gynäkologie, Vienna
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Denmark (2):
  - Herlev Hospital; Onkologisk afdeling, Herlev
  - Rigshospitalet, Onkologisk Klinik, København Ø
- France (10):
  - Institut Bergonie; Oncologie, Bordeaux
  - Centre Francois Baclesse; Oncologie, Caen
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - CRLCC Val dAurelle Paul Lam, Montpellier
  - Hopital Tenon; Oncologie Radiotherapie, Paris
  - Ch Lyon Sud; Chir Onc Gyne Sct Jules Courmont, Pierre-Bénite
  - Clinique Armoricaine Radiologie; Hopital de Jour, Plérin
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Centre Alexis Vautrin; Oncologie Medicale, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy; Oncologie Medicale, Villejuif
- Germany (19):
  - St. Elisabeth Krankenhaus Köln GmbH; Gynäkologie und Geburtshilfe, Cologne
  - Universitätsklinikum "Carl Gustav Carus"; Frauenheilkunde und Geburtshilfe, Dresden
  - Evangelischen Krankenhauses Düsseldorf; Frauenklinik, Düsseldorf
  - Universitätsklinikum Essen; Zentrum Für Frauenheilkunde, Essen
  - Kliniken Essen-Mitte Evang. Huyssens-Stiftung, Klinik für Gynäkologie und gynäkologische Onkologie, Essen
  - Universitätsklinikum Freiburg; Frauenklinik, Freiburg im Breisgau
  - Universitätsklinikum Greifswald; Klinik für Frauenheilkunde und Brustzentrum, Greifswald
  - Universitätsklinikum Hamburg-Eppendorf (UKE); Klinik und Poliklinik für Gynäkologie, Hamburg
  - Gynaekologisch-Onkologische Schwerpunktpraxis Prof. Dr. med. Lueck, Dr. Schrader und Dr. Noeding, Hanover
  - Nationales Centrum für Tumorerkrankungen (NCT) ; Gyn. Onk. Frauenklinik; Uniklinikum Heidelberg, Heidelberg
  - UNI-Klinikum Campus Kiel Klinik f.Gynäkologie u.Geburtshilfe, Kiel
  - Klinikum Konstanz, Frauenklinik, Konstanz
  - Klinikum rechts der Isar der TU München; Frauenklinik & Poliklinik, München
  - Sana Klinikum Offenbach GmbH; Klinik für Gynäkologie & Geburtshilfe, Offenbach
  - Hämatologisch/Onkologische Praxis Dr. Herbrick - Zipp/Prof. Dr. Decker, Studienzentrum, Ravensburg
  - Universitätsfrauen- und Poliklinik am Klinikum Suedstadt, Rostock
  - Universitätsklinik Tübingen; Frauenklinik, Tübingen
  - Universitätsklinikum Ulm Am Michelsberg; Frauenklinik, Ulm
  - HELIOS Dr. Horst Schmidt Kliniken Wiesbaden; Klinik für Gynäkologie und gynäkologische Onkologie, Wiesbaden
- Italy (7):
  - Istituto Tumori Napoli;Unità Operativa Oncologia Medica Uro-Ginecologica, Napoli, Campania
  - Istituto Regina Elena; Oncologia Medica A, Rome, Lazio
  - Ente Ospedaliero Ospedali Galliera; S.C. Oncologia Medica, Genoa, Liguria
  - A.O.Spedali Civili; Ostetricia e Ginecologia, Brescia, Lombardy
  - Istituto Nazionale dei Tumori; Divisione Oncologia Chirurgica e Ginecologica, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - A.O.U Pisana; Dipartimento di Ginecologia Oncologica, Pisa, Tuscany
- Netherlands (4):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Academ Ziekenhuis Groningen; Medical Oncology, Groningen
  - Academisch Ziekenhuis Leiden; Clinical Oncology, Leiden
  - UMC St Radboud, Nijmegen
- The Norvegian Radium Hospital Montebello; Dept of Oncology, Oslo, Norway
- Spain (20):
  - Hospital Son Llatzer; Servicio de Oncologia, Palma de Mallorca, Balearic Islands
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona, Barcelona
  - Hospital Duran i Reynals; Oncologia, Barcelona, Barcelona
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Barcelona, Barcelona
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Hospital Universitari de Girona Dr. Josep Trueta; Servicio de Oncologia, Girona, Girona
  - Hospital Universitari Arnau de Vilanova de Lleida; Servicio de Oncologia, Lleida, Lerida
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid, Madrid
  - Centro Oncologico MD Anderson Internacional; Servicio de Oncologia, Madrid, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC); Dirección Médica, Madrid, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Oncologia, Málaga, Malaga
  - Hospital Universitario Virgen de Arrixaca; Servicio de Oncologia, Murcia, Murcia
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia, Valencia
  - Hospital Universitario la Fe; Servicio de Oncologia, Valencia, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza, Zaragoza
- Sweden (2):
  - Universitetssjukhuset; Onkologkliniken, Linköping
  - Skånes University Hospital, Skånes Department of Onclology, Lund

REFERENCES:
- [Derived] Lorusso D, Hilpert F, Gonzalez Martin A, Rau J, Ottevanger P, Greimel E, Luck HJ, Selle F, Colombo N, Kroep JR, Mirza MR, Berger R, Pardo B, Grischke EM, Berton-Rigaud D, Martinez-Garcia J, Vergote I, Redondo A, Cardona A, Bastiere-Truchot L, du Bois A, Kurzeder C; PENELOPE trial investigators. Patient-reported outcomes and final overall survival results from the randomized phase 3 PENELOPE trial evaluating pertuzumab in low tumor human epidermal growth factor receptor 3 (HER3) mRNA-expressing platinum-resistant ovarian cancer. Int J Gynecol Cancer. 2019 Sep;29(7):1141-1147. doi: 10.1136/ijgc-2019-000370. Epub 2019 Aug 15. PMID 31420414

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 208 participants were entered into the study, 52 participants in Part 1, and 156 participants in Part 2 of the study. Of these, 203 received treatment with pertuzumab or pertuzumab-placebo (50 participants in Part 1 and 153 participants in Part 2).
Groups:
- Part 2: Placebo+Chemotherapy: Participants received pertuzumab-matching placebo and chemotherapy (paclitaxel or topotecan or gemcitabine) in cycles of 3 weeks until progressive disease as per investigator's assessment, unacceptable toxicity, withdrawal of consent, or death. Chemotherapy was administered as per investigators discretion.
Period: Part 1: Safety Run in Phase
Arm/Group | Part 1: Pertuzumab + Topotecan | Part 1: Pertuzumab + Paclitaxel | Part 2: Pertuzumab+Chemotherapy | Part 2: Placebo+Chemotherapy
Started | 22 | 28 | 0 | 0
Completed | 6 | 5 | 0 | 0
Not Completed | 16 | 23 | 0 | 0
Not completed — Participants withdrawn consent | 1 | 1 | 0 | 0
Not completed — Death | 15 | 20 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Period: Part 2: Randomized Phase
Arm/Group | Part 1: Pertuzumab + Topotecan | Part 1: Pertuzumab + Paclitaxel | Part 2: Pertuzumab+Chemotherapy | Part 2: Placebo+Chemotherapy
Started | 0 | 0 | 78 | 78
Participants Randomized But Not Treated | 0 | 0 | 1 | 2
Participants Mis-randomized | 0 | 0 | 2 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 78 | 78
Not completed — Participant withdrew consent | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 62 | 68
Not completed — Alive at data-cut | 0 | 0 | 13 | 7
Not completed — Participant noncompliance | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Part 1: all participants enrolled and treated in Part 1 of the study ('as treated' analysis) and Part 2: intent-to-treat (ITT) population was defined as all randomized participants in the group to which they were randomly assigned ('as randomized' analysis).
Groups:
- Part 1: Pertuzumab + Topotecan: Participants received pertuzumab and topotecan in cycles of 3 weeks until progressive disease as per investigators assessment, unacceptable toxicity, withdrawal of consent, or death.
- Part 1: Pertuzumab + Paclitaxel: Participants received pertuzumab and paclitaxel in cycles of 3 weeks until progressive disease as per investigators assessment, unacceptable toxicity, withdrawal of consent, or death.
- Part 2: Pertuzumab+Chemotherapy: Participants received pertuzumab and chemotherapy (paclitaxel or topotecan or gemcitabine) in cycles of 3 weeks until progressive disease as per investigators assessment, unacceptable toxicity, withdrawal of consent, or death. Chemotherapy was administered as per investigators discretion.
- Part 2: Placebo+Chemotherapy: Participants received pertuzumab matching placebo and chemotherapy (paclitaxel or topotecan or gemcitabine) in cycles of 3 weeks until progressive disease as per investigators assessment, unacceptable toxicity, withdrawal of consent, or death. Chemotherapy was administered as per investigators discretion.
- Total: Total of all reporting groups
Arm/Group | Part 1: Pertuzumab + Topotecan | Part 1: Pertuzumab + Paclitaxel | Part 2: Pertuzumab+Chemotherapy | Part 2: Placebo+Chemotherapy | Total
Number analyzed (Participants) | 22 | 28 | 78 | 78 | 206
Age, Customized [Number; unit: participants]
  Less than or equal to (≤)65 years | 15 | 17 | 40 | 44 | 116
  Greater than (>)65 years | 7 | 11 | 38 | 34 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 78 | 78 | 206
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants With Adverse Events (AEs)
Description: An AE can be any unfavorable and unintended sign (including an abnormality laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Approximately 28 months (assessed at screening, baseline until 28 days after the last dose of study treatment)
Population: All Treated population included all participants enrolled and treated in Part 1 of the study ('as treated' analysis) and who had received at least 1 dose of pertuzumab or chemotherapy.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Pertuzumab + Topotecan | Part 1: Pertuzumab + Paclitaxel
Number analyzed (Participants) | 22 | 28
percentage of participants | 95.5 | 100.0

2. Primary Outcome: Part 2: Progression Free Survival (PFS) as Assessed by a Blinded Independent Review Committee (IRC) Including Malignant Bowel Obstruction (MBO)
Description: PFS (IRC-Assessed) was defined as the time from randomization into Part 2 of the trial until progressive disease (PD), MBO or death from any cause, whichever occurred first per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. PD could base on symptom deterioration or was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of one or more new lesions and/or the unequivocal progression of existing non-target lesions.
Time Frame: Approximately 44 months (assessed at screening and every 9 weeks from randomization until disease progression)
Population: ITT Population was defined as all randomized participants in the group to which they were randomly assigned ('as randomized' analysis).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Pertuzumab+Chemotherapy | Part 2: Placebo+Chemotherapy
Number analyzed (Participants) | 78 | 78
months | 4.27 [3.65 to 6.11] | 2.74 [2.14 to 4.73]
Statistical Analysis 1: Comparison: Part 2: Pertuzumab+Chemotherapy vs Part 2: Placebo+Chemotherapy; The stratified time-to-event analysis included the treatment group variable plus the following stratification factors: selected chemotherapy cohort (gemcitabine versus topotecan vs paclitaxel), previous anti-angiogenic therapy (yes versus no), and progression-free interval (PFI) since platinum therapy (< 3 months versus 3-6 months). A hazard ratio < 1 favored the pertuzumab + chemotherapy treatment arm; Test type: Superiority or Other; p = 0.4983, 2 sided log-rank; Hazard Ratio (stratified) = 0.88, 95% CI 2-sided [0.62 to 1.27]

3. Secondary Outcome: Part 1- Objective Response Rate (ORR)
Description: ORR was defined as the number of participants with best overall response (BOR) of complete response (CR) or partial response (PR) recorded from the start of treatment, until the end of treatment. BOR documented as confirmed CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeter (mm). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Approximately 28 months (assessed at baseline and every 9 weeks from randomization until disease progression)
Population: All Treated participants with measurable disease at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Pertuzumab + Topotecan | Part 1: Pertuzumab + Paclitaxel
Number analyzed (Participants) | 14 | 24
percentage of participants | 14.3 | 25.0

4. Secondary Outcome: Part 2- Objective Response Rate (ORR)
Description: ORR was defined as the number of participants with BOR of CR or PR recorded from the start of treatment, until the end of treatment. BOR documented as confirmed CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeter (mm). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Approximately 44 months (assessed at screening and every 9 weeks from randomization until disease progression)
Population: ITT population with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Pertuzumab+Chemotherapy | Part 2: Placebo+Chemotherapy
Number analyzed (Participants) | 61 | 69
percentage of participants | 14.8 [7.0 to 26.2] | 8.7 [3.3 to 18.0]
Statistical Analysis 1: Comparison: Part 2: Pertuzumab+Chemotherapy vs Part 2: Placebo+Chemotherapy; Test type: Superiority or Other; p = 0.4102, Fisher Exact; Difference in response rate = 6.06, 95% CI 2-sided [6.0 to 18.3] — Approximate 95% CI for difference of 2 rates using Hauck-Anderson method

5. Secondary Outcome: Part 1: PFS Assessed by the Investigator
Description: PFS as assessed by Investigator was defined as the time from first dose of pertuzumab or chemotherapy in Part 1 of the trial, until disease progression according to RECIST version 1.1, symptomatic deterioration or death from any cause, whichever occurs first. PD could base on symptom deterioration or was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of one or more new lesions and/or the unequivocal progression of existing non-target lesions. Participants were censored at the last tumor assessment. Participants who have no tumor assessments after baseline and who were still alive will be censored at 1 day.
Time Frame: Approximately 28 months (assessed at screening and every 9 weeks from randomization until disease progression)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Pertuzumab + Topotecan | Part 1: Pertuzumab + Paclitaxel
Number analyzed (Participants) | 22 | 28
months | 4.07 [1.94 to 6.08] | 4.24 [3.45 to 6.01]

6. Secondary Outcome: Part 2: Progression-free Survival (PFS) Assessed by the Investigator
Description: PFS (Investigator-assessed) is defined as the time from randomization, until disease progression according to RECIST v1.1 including death or MBO, whichever occurs first. Censoring is based on the last tumor assessment. If no tumor assessment post baseline, then censoring is at day 1. PD could base on symptom deterioration or was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of one or more new lesions and/or the unequivocal progression of existing non-target lesions.
Time Frame: Approximately 44 months (assessed at screening and every 9 weeks from randomization until disease progression)
Population: ITT Population included all randomized participants in the group to which they were randomly assigned ('as randomized' analysis)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Pertuzumab+Chemotherapy | Part 2: Placebo+Chemotherapy
Number analyzed (Participants) | 78 | 78
months | 4.22 [3.25 to 5.22] | 3.94 [2.63 to 4.30]

7. Secondary Outcome: Part 2: European Organization for Research and Treatment of Cancer (EORTC) Quality of Life (QoL) Questionnaire (QLQ) of Core 30 (C30) Score
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4-point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale [1 'very poor' to 7 'Excellent']). Scores averaged, transformed to 0-100 scale; for functional scores, a higher score represents a better level of functioning. For symptom scores, a higher score represents a more severe level of symptoms. For the global health status scores, a higher score represents a better quality of life.
Time Frame: Baseline (assessed at baseline and every 9 weeks from randomization until disease progression)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 2: Pertuzumab+Chemotherapy | Part 2: Placebo+Chemotherapy
Number analyzed (Participants) | 78 | 78
units on a scale
  Functional Scales: Physical (n=71, 74) | 71.1 (22.77) | 74.9 (20.85)
  Functional Scales: Role (n=70, 73) | 68.6 (33.16) | 69.4 (32.40)
  Functional Scales: Emotional (n=71, 73) | 59.5 (24.03) | 65.9 (23.42)
  Functional Scales: Cognitive (n=71, 73) | 81.2 (25.34) | 84.9 (20.25)
  Functional Scales: Social (n=71, 73) | 70.7 (30.01) | 68.3 (29.81)
  Symptomatic Scales: Fatigue (n=71, 74) | 41.2 (28.75) | 38.4 (27.77)
  Symptomatic Scales: Nausea and vomiting (n=72, 74) | 10.4 (15.68) | 12.4 (20.47)
  Symptomatic Scales: Pain (n=72, 74) | 35.2 (31.34) | 31.1 (29.24)
  Symptomatic Scales: Dyspnoea (n=68, 73) | 22.5 (28.47) | 21.5 (27.98)
  Symptomatic Scales: Insomnia (n=69, 74) | 35.3 (31.25) | 31.5 (31.16)
  Symptomatic Scales: Appetite loss (n=71, 73) | 24.9 (30.19) | 21.0 (26.36)
  Symptomatic Scales: Constipation (n=69, 72) | 25.6 (32.41) | 26.4 (32.59)
  Symptomatic Scales: Diarrhoea (n=69, 72) | 14.5 (26.49) | 14.4 (22.26)
  Symptomatic Scales:Financial difficulties(n=70,72 | 17.6 (28.78) | 13.4 (22.83)
  Global health status / QoL scale (n=71, 72) | 54.1 (24.99) | 61.1 (22.29)

8. Secondary Outcome: Part 2: Percentage of Participants With Adverse Events (AEs)
Description: as for outcome 1
Time Frame: Approximately 28 months (assessed at screening, baseline until 28 days after the last dose of study treatment)
Population: Safety population included all participants who had received at least 1 dose of pertuzumab, pertuzumab-placebo, or chemotherapy.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Pertuzumab+Chemotherapy | Part 2: Placebo+Chemotherapy
Number analyzed (Participants) | 77 | 76
percentage of participants | 98.7 | 100

9. Secondary Outcome: Part 2: Overall Survival
Description: Overall survival was defined as the time from randomization into Part 2 of the trial until death from any cause
Time Frame: Approximately 44 months (assessed at screening and every 9 weeks from randomization until disease progression)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Pertuzumab+Chemotherapy | Part 2: Placebo+Chemotherapy
Number analyzed (Participants) | 78 | 78
months | 10.18 [6.67 to 15.24] | 8.36 [6.14 to 11.99]
Statistical Analysis 1: Comparison: Part 2: Pertuzumab+Chemotherapy vs Part 2: Placebo+Chemotherapy; The stratified time-to-event analysis included the treatment group variable plus the following stratification factors: selected chemotherapy cohort (gemcitabine versus topotecan versus paclitaxel), previous angiogenic therapy (yes versus no) and PFI since platinum therapy (<3 months versus 3-6 months); Test type: Superiority or Other; p = 0.5960, 2 sided log-rank; Hazard ratio (stratified) = 0.90, 95% CI 2-sided [0.61 to 1.32] — A hazard ratio < 1 favored the Pertuzumab + Chemotherapy treatment group

ADVERSE EVENTS:
Time Frame: Approximately 28 months (assessed at screening, baseline until 28 days after the last dose of study treatment)
Arm/Group | Part 1: Pertuzumab + Topotecan | Part 1: Pertuzumab + Paclitaxel | Part 2: Pertuzumab+Chemotherapy | Part 2: Placebo+Chemotherapy
Serious Adverse Events (participants affected / at risk) | 9/22 | 11/28 | 29/77 | 33/76
Other Adverse Events (participants affected / at risk) | 21/22 | 27/28 | 72/77 | 75/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Pertuzumab + Topotecan (N=22) | Part 1: Pertuzumab + Paclitaxel (N=28) | Part 2: Pertuzumab+Chemotherapy (N=77) | Part 2: Placebo+Chemotherapy (N=76)
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 4
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 4 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Subileus (Gastrointestinal disorders) | 1 | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1
Abdominal Infection (Infections and infestations) | 0 | 1 | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 1 | 1
Pyrexia (General disorders) | 0 | 2 | 1 | 2
Death (General disorders) | 0 | 1 | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Bone Marrow Failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 2 | 3
Performance Status Decreased (General disorders) | 0 | 0 | 0 | 1
Anal Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 1
Infective Myositis (Infections and infestations) | 0 | 0 | 1 | 0
Kidney Infection (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis Pneumococcal (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Contrast Media Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 2 | 1
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 1
Weight Decreased (Investigations) | 0 | 0 | 1 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 2
Cerebral Ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary Tract Disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Vaginal Fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 2
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Not yet coded (General disorders) | 0 | 0 | 1 | 0 — This adverse event was not coded at the time of the primary analysis. The preferred term will be reported when available at the final analysis.
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Pertuzumab + Topotecan (N=22) | Part 1: Pertuzumab + Paclitaxel (N=28) | Part 2: Pertuzumab+Chemotherapy (N=77) | Part 2: Placebo+Chemotherapy (N=76)
Diarrhoea (Gastrointestinal disorders) | 14 | 22 | 50 | 23
Nausea (Gastrointestinal disorders) | 11 | 10 | 31 | 34
Vomiting (Gastrointestinal disorders) | 13 | 5 | 19 | 23
Abdominal Pain (Gastrointestinal disorders) | 6 | 4 | 16 | 21
Constipation (Gastrointestinal disorders) | 5 | 5 | 12 | 22
Stomatitis (Gastrointestinal disorders) | 2 | 5 | 9 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 1 | 6 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 4 | 3
Dry Mouth (Gastrointestinal disorders) | 0 | 2 | 2 | 7
Rectal Haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Asthenia (General disorders) | 14 | 8 | 32 | 24
Fatigue (General disorders) | 5 | 10 | 21 | 24
Pyrexia (General disorders) | 5 | 5 | 9 | 12
Mucosal Inflammation (General disorders) | 7 | 2 | 11 | 6
Oedema Peripheral (General disorders) | 5 | 2 | 12 | 9
Influenza Like Illness (General disorders) | 3 | 0 | 4 | 1
Malaise (General disorders) | 0 | 2 | 0 | 0
Oedema (General disorders) | 0 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 15 | 10 | 28 | 32
Neutropenia (Blood and lymphatic system disorders) | 5 | 3 | 23 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 3 | 5
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 4 | 9
Thrombocytosis (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 10 | 15 | 21
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 3 | 4 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 3 | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 7 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 7 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Pain Of Skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 8 | 5 | 13 | 17
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 4 | 7 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 9 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 7 | 10 | 9
Headache (Nervous system disorders) | 3 | 1 | 7 | 5
Dizziness (Nervous system disorders) | 2 | 1 | 7 | 4
Neuropathy Peripheral (Nervous system disorders) | 1 | 2 | 7 | 9
Paraesthesia (Nervous system disorders) | 1 | 2 | 4 | 4
Ageusia (Nervous system disorders) | 0 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 9 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 16 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 7 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 7 | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 6 | 8 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4 | 5
Nasopharyngitis (Infections and infestations) | 2 | 2 | 10 | 6
Urinary Tract Infection (Infections and infestations) | 3 | 1 | 7 | 4
Nail Infection (Infections and infestations) | 2 | 0 | 0 | 0
Weight Decreased (Investigations) | 2 | 2 | 2 | 4
Ejection Fraction Decreased (Investigations) | 0 | 2 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 5 | 5
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 2 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 4 | 5
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 4 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 5 | 6
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 6 | 5
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 3 | 7
Neutrophil Count Decreased (Investigations) | 0 | 0 | 7 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 3 | 5
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 3 | 5
Platelet Count Decreased (Investigations) | 0 | 0 | 6 | 2
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 4
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 4 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 4 | 1
Hypertension (Vascular disorders) | 0 | 0 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.